CLINICAL TRIAL: NCT06652711
Title: Addressing the Mental Health and Emotional Well-being of Immigrants Through a Scalable Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005337
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-06

CONDITIONS: Well-being; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- 2-month access and no incentive (Experimental): Participants have access to the well-being app for two months and receive no incentive for using the app.
  Interventions: Behavioral: 2-month access to mental health app
- 2-month access and lottery incentive (Experimental): Participants have access to the well-being app for two months, and participate in a lottery for gift cards if they display sufficient engagement.
  Interventions: Behavioral: 2-month access to mental health app; Behavioral: Lottery incentive
- 2-month access and direct incentive (Experimental): Participants have access to the well-being app for two months, and receive a direct payment if they display sufficient engagement.
  Interventions: Behavioral: 2-month access to mental health app; Behavioral: Direct incentive
- 4-month access and no incentive (Experimental): Participants have access to the well-being app for four months and receive no incentive for using the app.
  Interventions: Behavioral: 4-month access to mental health app
- 4-month access and lottery incentive (Experimental): Participants have access to the well-being app for four months, and participate in a lottery for gift cards if they display sufficient engagement.
  Interventions: Behavioral: 4-month access to mental health app; Behavioral: Lottery incentive
- 4-month access and direct incentive (Experimental): Participants have access to the well-being app for four months, and receive a direct payment if they display sufficient engagement.
  Interventions: Behavioral: Direct incentive; Behavioral: 4-month access to mental health app
- control (No Intervention): Participants do not have access to the app during the study.

INTERVENTIONS:
Behavioral: 2-month access to mental health app — Participants will have access to the well-being app for two months.
  Arms: 2-month access and direct incentive; 2-month access and lottery incentive; 2-month access and no incentive
Behavioral: Direct incentive — A $10 gift card are given to participants at the end of the study if they used the app sufficiently.
  Arms: 2-month access and direct incentive; 4-month access and direct incentive
Behavioral: 4-month access to mental health app — Participants will have access to the well-being app for four months.
  Arms: 4-month access and direct incentive; 4-month access and lottery incentive; 4-month access and no incentive
Behavioral: Lottery incentive — Participants can participate in a draw of $150 gift cards at the end of the study if they used the app sufficiently.
  Arms: 2-month access and lottery incentive; 4-month access and lottery incentive

SUMMARY:
We will study the impacts of offering access to an emotional well-being phone app to Hispanic U.S. immigrants in psychological distress. Our primary outcome is participants' psychological well-being.

ELIGIBILITY:
The target population will be: immigrants to the U.S. of Hispanic origin whose native language is Spanish, who have been living in the U.S. (intermittently or continuously) for less than 10 years, who are over 18 years of age, who have a PHQ4 score that is three or more, who would be interested in using a well-being phone app, who do not have a graduate degree and have access to a smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Depression, anxiety, and stress | Up to six months since enrollment
  Measured by the Patient Health Questionnaire 8 (PHQ)
Anxiety | Up to six months since enrollment
  Measured by GAD-7 (General Anxiety Disorder Questionnaire)
Stress | Up to six months since enrollment
  Measured by PSS-4 (Perceived Stress Scale 4)
Self-efficacy | Up to six months since enrollment
  Measured using the short version of the General Self-Efficacy Scale, the GSE-6
Locus of Control | Up to six months since enrollment
  Measure using the Internal-External Locus of Control Short Scale-4 (IE-4)

SECONDARY OUTCOMES:
Remittances | Up to six months since enrollment
  Amount and frequency of remittances to the participants' countries of origin
Social connectedness and Integration to the US | Up to six months since enrollment
  we will measure this with a subset of questions of the Multidimensional Measure of Immigrant Integration (Harder et al. 2018), with questions about: psychological integration, linguistic integration, political and economic integration and social integration. We will report these separately and combining them through an Anderson index (Anderson, 2008). In addition, as a second outcome we will use a revealed-choice measures of their demand to invest in learning English (by giving them a choice between access to a language course or cash/item)

OTHER OUTCOMES:
Perceptions and attitudes towards using mental health services | Up to six months since enrollment
  Provided that there was widespread reticence at baseline.
Parental expectations and aspirations about their youngest child under 18 educational attainment | Up to six months since enrollment
  For those with children
Absenteeism | Up to six months since enrollment
  Question about missing day at work in the last month
Uptake for the app | Up to six months since enrollment
  Number of participants who download the app
Use of the app | Up to six months since enrollment
  Number of days and minutes participants use the app
Demand for the app | Up to six months since enrollment
  Willingness to pay exercise to recover demand for the app

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No